CLINICAL TRIAL: NCT02846740
Title: Cranial Electric Stimulation to Modify Suicide Risk Factors in Psychiatric Inpatients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No finding at halfway point of the study
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Nithin Krishna, Assistant Professor of Psychiatry, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00065640
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Suicide; Depression; Anxiety; Insomnia; Agitation
Keywords: cranial electric stimulation; suicide; psychiatric inpatients
MeSH Terms: conditions — Suicide; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Adjunctive CES (Experimental): CES 100µA for one hour daily, five to seven days per week. Rating scales will be administered at baseline (i.e., pre-treatment), twice a week and at the end of the study.
  Interventions: Device: Alpha-Stim®.; Behavioral: Montgomery-Åsberg Depression Rating Scale, Hamilton Anxiety Rating Scale, The Pittsburgh Sleep Quality Index and agitated behavior Scale
- Sham control CES (Sham Comparator): For the sham group the Alpha-Stim® will not emit electricity. All other procedures will be the same for both the sham group and the active CES group. The current intensity will be preset and locked by the manufacturer. The sham devices will appear identical to the active device.
  Interventions: Device: Alpha-Stim®.; Behavioral: Montgomery-Åsberg Depression Rating Scale, Hamilton Anxiety Rating Scale, The Pittsburgh Sleep Quality Index and agitated behavior Scale

INTERVENTIONS:
Device: Alpha-Stim®. — cranial electrical stimulation
Behavioral: Montgomery-Åsberg Depression Rating Scale, Hamilton Anxiety Rating Scale, The Pittsburgh Sleep Quality Index and agitated behavior Scale — A summed global score from rating scales measuring the Modifiable suicide risk factors (MSRF's).

SUMMARY:
This pilot study aims to investigate whether a treatment called cranial electric stimulation or CES can decrease risk factors for suicide. The specific CES device we will use is called Alpha-Stim®. CES will be used in addition to usual treatment (medication and group therapy).

DETAILED DESCRIPTION:
Suicide is still a major issue in the United States and all around the world. There are many reasons for people attempting suicide and the major modifiable risk factors are depression, anxiety, insomnia, and agitation. The standard treatment for all suicidal patients includes medication, admission to a hospital and reducing the risk factors. Medications have potential side effects and concerns about the drug interactions. One of the biological treatment alternatives to medication is cranial electric stimulation. This technique uses a device to stimulate the brain through electrical current. Using an Alpha-Stim® device, current is applied to the brain using skin electrodes which can be easily clipped on to the earlobe. The amount of current used is very low and is 1/1000 th of the current used for electroconvulsive therapy (ECT) and 1/10 th to 1/20 th of the 1-2 milliamperes used with transcranial direct current stimulation (tDCS). Our goal is to examine the safety and efficacy of this device when used as an add-on or adjunctive treatment to the usual treatments during the inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a patient admitted voluntarily to the UMMC adult psychiatric inpatient services with suicidal thoughts / intent / plan or suicide attempt who also has MSRFs including anxiety, agitation, insomnia, and/or depression).
2. Subject must be between the ages of 18 and 65 (inclusive). Both men and women will be included
3. Subjects who are female must have a negative pregnancy test prior to enrolling in the study, and must be practicing at least one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, or oral/hormonal contraception or abstinence, which is typically the case on the inpatient units.
4. If a subject has a substance abuse disorder, they must also have another non-substance abuse psychiatric disorder as determined from the clinical history.
5. Chronic medical conditions such as endocrine disease, hypertension, renal disease, must be stable.
6. Subject must be capable of giving informed consent. Subject must provide written informed consent prior to study participation.
7. Subject must be capable of doing active or sham CES treatments and completing all study requirements.

Exclusion Criteria:

1. Subject has a significant medical disorder with acute symptoms which could impair reliable participation in the trial or affect their MSRFs.
2. Subject is pregnant.
3. Subject has had concomitant therapy with another investigational drug, or participation in an investigational drug study within one month prior to entering this study.
4. Subject has a clinical history of poor compliance or in the investigator's judgment participation in the study would be clinically contraindicated.
5. Subject has current or past behavior that suggests to the investigator that his/her suicidal behavior is driven by secondary gain, i.e. expressing suicidal thoughts so that s/he can be admitted due to homelessness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nithin E Krishna, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjunctive CES | Sham Control CES
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjunctive CES | Sham Control CES | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.87 (2) | 31.87 (2.5) | 32.87 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Modifiable Suicide Risk Factors (MSRF's) Global Score
Description: Efficacy of adjunctive cranial electric stimulation (CES), specifically Alpha-Stim®, to reduce suicide risk in psychiatric inpatients through a randomized, double-blind, sham-controlled, clinical trial. The primary efficacy outcome measure will be change in the modifiable suicide risk factors (MSRF's) as indicated by a summed global score from rating scales measuring the MSRFs that include Montgomery-Åsberg Depression Rating Scale (range very severe = 44; severe = 31; moderate = 25; mild = 15; & recovered = 7), Hamilton Anxiety Rating Scale (range of 0-56, <17 indicates mild severity, 18-24, moderate severity & 25-30 severe). Both scales were summed, the full theoretical scale range is 0-116, with higher scores indicating a worse outcome. Due to short hospital stays, we were not able to use Agitated Behavior Scale and Pittsburgh Sleep Quality Index scale in a meaningful manner to include in our analysis, so we did not include that scale.
Time Frame: Baseline, 22 months,
Population: Many patients were discharged within a few days of admission, some left in two days, which left us with just baseline and several missing scales.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adjunctive CES | Sham Control CES
Number analyzed (Participants) | 15 | 15
score on a scale | 35.33 (1.02) | 36.5 (1.04)

2. Primary Outcome: Adverse Effects and Safety
Description: Safety of adjunctive cranial electric stimulation (CES), specifically Alpha-Stim®, to reduce suicide risk in psychiatric inpatients through a randomized, double-blind, sham-controlled, clinical trial. The primary safety outcome measure will be responses to an adverse effect assessment questionnaire (GASE questionnaire).
Time Frame: Baseline, 22 months,
Measure: Count of Participants; unit: Participants
Arm/Group | Adjunctive CES | Sham Control CES
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

3. Secondary Outcome: Length of Stay
Time Frame: Baseline, 22 months,
Population: This was a difficult analysis considering patients had different motives for staying versus discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Adjunctive CES | Sham Control CES
Number analyzed (Participants) | 15 | 15
Days | 11 (0.5) | 12 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study, up to 22 months.
Description: There were no reports of any serious adverse events or side effects from due to the study.
Arm/Group | Adjunctive CES | Sham Control CES
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT02846740/SAP_000.pdf
  • Informed Consent Form (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT02846740/ICF_001.pdf
  • Study Protocol (2016-02-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02846740/Prot_002.pdf